CLINICAL TRIAL: NCT05744648
Title: Clinical Efficacy of a Novel Titania Nanoparticle-Reinforced Bonding Agent in Reducing Post-Restorative Sensitivity: A Randomized Clinical Trial
Brief Title: Efficacy of Nanoparticle-incorporated Bonding Agent on Post-restorative Sensitivity
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Pakistan Institute of Medical Sciences (Other Government)
Responsible Party: Principal Investigator, NEHAL AMIR, Principal Investigator, Pakistan Institute of Medical Sciences
Allocation: Non-Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: SOD/ERB/2022/14
Record Dates: First submitted 2023-02-16; First posted 2023-02-27 (Actual); Last update posted 2023-09-13 (Actual); Status verified 2023-09

CONDITIONS: Carious Lesion
Keywords: Composite resins; Dentin bonding agents; Dentin Sensitivity; Nanoparticles; Titania
MeSH Terms: conditions — Dental Caries; Dentin Sensitivity

STUDY DESIGN:
Intervention Model Description: In this study, participants will be allocated in two groups by Consecutive non-random sampling technique.
Who Masked: Participant, Care Provider, Outcomes Assessor
Masking Description: This is a triple-blinded study in which the participant, care provider and outcome assessor will be masked.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Group A (Experimental): Group A will receive composite resin restoration with Titania nanoparticle incorporated bonding agent
  Interventions: Procedure: Composite resin restoration using Titania nanoparticle reinforced bonding agent
- Group B (Experimental): Group B will receive composite resin restoration without Titania nanoparticle incorporated bonding agent
  Interventions: Procedure: Composite resin restoration without Titania nanoparticle incorporated bonding agent

INTERVENTIONS:
Procedure: Composite resin restoration using Titania nanoparticle reinforced bonding agent — Each group will receive Composite resin restoration for Class-I and Class-II carious lesion. In group A, titania nanoparticle reinforced bonding agent will be used
  Arms: Group A
Procedure: Composite resin restoration without Titania nanoparticle incorporated bonding agent — Composite resin restoration without Titania nanoparticle incorporated bonding agent
  Arms: Group B

SUMMARY:
Type of study: Randomized Clinical trial To compare post-restorative sensitivity between titania nanoparticle reinforced bonding agent and bonding agent without nanoparticles in posterior composite restorations.

Participants aged 18 years and above with Class-I and Class-II Carious lesions are allocated in two groups. Group A will undergo composite restoration with Nanoparticles incorporated in bonding agent. Group B will undergo restoration without nanoparticles in bonding agent.

DETAILED DESCRIPTION:
In this study Novel titania nanoparticle reinforced bonding agent will be evaluated for post-restorative sensitivity in composite restorations. Participants following the Inclusion criteria will be allocated in this study by Consecutive non-random sampling technique. Participants will be divided into two groups A and B. After rubber dam isolation, carious lesion will be excavated. In group A, titania nanoparticle reinforced bonding agent will be used for restorative treatment while in group B, Bonding agent without nanoparticles will be used. Post-restorative sensitivity record will be taken at 24 hours, after one week and after one month. Sensitivity will be assessed using Visual analog scale (VAS) mean score.

ELIGIBILITY:
Inclusion Criteria:

* Participants with good general health
* Selected teeth should be vital and periodontally healthy
* Class-I and II with minimal cavity depth of 3mm, not exceeding 5mm
* Defective previous restorations in need of replacement (secondary caries/fractures)
* Selected teeth should be in occlusion with natural or prosthetic antagonist and adjacent teeth

Exclusion Criteria:

* Patients with Temporomandibular disorders
* Extremely poor oral hygiene status
* Teeth with very deep carious lesions
* Teeth with periapical or periodontal pathology
* Patients taking anti-inflammatory, analgesics or psychotropic drugs
* History of spontaneous pain
* Previously root canal treated teeth

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2023-01-05 (Actual); Primary Completion 2023-06-20 (Actual); Study Completion 2023-06-20 (Actual)

PRIMARY OUTCOMES:
Post-restorative sensitivity in composite resin restoration | 1 month
  Evaluation of bonding agent with titania nanoparticles and without nanoparticles on post-restorative sensitivity using Visual analog scale with scoring from 0 to 10. Score 10 means worst outcomes

CONTACTS AND LOCATIONS:
Overall Officials: Nehal Amir, BDS, Principal Investigator — Pakistan Institute of Medical Sciences
Locations (1):
- School of Dentistry, Pakistan Institute of Medical Sciences, Islamabad, Pakistan

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Aboelenein AZ, Riad MI, Haridy MF. Effect of a Self-Etch Adhesive Containing Nanobioglass on Postoperative Sensitivity of Posterior Composite Restorations - A Randomized Trial. Open Access Maced J Med Sci. 2019 Jul 25;7(14):2313-2320. doi: 10.3889/oamjms.2019.585. eCollection 2019 Jul 30. PMID 31592280
- [Background] Melo MA, Cheng L, Zhang K, Weir MD, Rodrigues LK, Xu HH. Novel dental adhesives containing nanoparticles of silver and amorphous calcium phosphate. Dent Mater. 2013 Feb;29(2):199-210. doi: 10.1016/j.dental.2012.10.005. Epub 2012 Nov 6. PMID 23138046